CLINICAL TRIAL: NCT07150494
Title: Predictive and Diagnostic Value of BIND Score in Assessment of Severe Neonatal Jaundice Cases in NICU
Brief Title: Predictive and Diagnostic Value of BIND Score in Assessment of Severe Neonatal Jaundice Cases in Neonatal Intensive Care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nouralhoda Ahmed Metwally Ibrahim, Nouralhoda Ahmed, Assiut University
Other Study IDs: Neonatal jaundice cases in nic
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Phototherapy — Phototherapy used to decrease high billirubin level in neonatal jaundice

SUMMARY:
Early detection and prevention of neonatal encephalopathy using BIND score.

ELIGIBILITY:
Inclusion criteria:

Newborn < 28 days old Neonates with severe hyperbilirubinemia need extensive phototherapy impending exchange transfusion

Exclusion criteria:

Age > 28 days old Neonates with any abnormal neurological signs suggesting neurological disease (hypoxic ischemic encephalopathy, muscle disease, …etc.).

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: Neonates with severe neonatal jaundice
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Decrease high billirubin level | One year duration
  We use bind score to evaluate neurological condition of neoborns then use photo therapy to decrease
Predictive and diagnostic value of BIND score in assessment of severe neonatal jaundice cases in NICU | Baseline
  Early detection and prevention of neonatal encephalopathy using BIND score.
Predictive and diagnostic value of BIND score in assessment of severe neonatal jaundice cases in NICU | Baseline

REFERENCES:
- [Background] Vongbhavit K, Rearkyai S, Janyoungsak P, Panburana J. Impact of 2022 AAP Neonatal Hyperbilirubinemia Guidelines in a Middle-Income Country: A Single-Center Study in Thailand. Neonatology. 2025;122(6):660-668. doi: 10.1159/000547630. Epub 2025 Aug 13. PMID 40815110
- See also: Related Info — https://bmcpediatr.biomedcentral.com/articles/10.1186/s12887-015-0355-2